CLINICAL TRIAL: NCT05166421
Title: Phase 1, Randomized, Open Label, Three-arm, Single Dose, Parallel Group Study to Compare AZD7442 (AZD8895 + AZD1061) Pharmacokinetic Exposure Following Intramuscular Administration as a Co-formulation Versus Administration From Two Separate Vials of the Individual Monoclonal Antibodies in Adult Healthy Participants
Brief Title: Study to Evaluate Pharmacokinetic Comparability Between AZD7442 Co-formulation (AZD8895 + AZD1061) vs AZD8895 and AZD1061 Individually in Adult Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8850C00009
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Corona Virus Disease
Keywords: Monoclonal antibodies; Adult healthy participants
MeSH Terms: interventions — cilgavimab and tixagevimab drug combination; tixagevimab; cilgavimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AZD7442 (co-formulation) (Experimental): Participants will receive single dose of AZD7442 (co-formulation of AZD8895 + AZD1061) on Day 1.
  Interventions: Biological: AZD7442
- AZD8895 and AZD1061 (clonal cell line material) (Active Comparator): Participants will receive two separate doses of the individual mAbs (AZD8895 and then AZD1061) on Day 1.
  Interventions: Biological: AZD8895 (clonal cell line material); Biological: AZD1061 (clonal cell line material)
- AZD8895 and AZD1061 (cell pool material) (Active Comparator): Participants will receive two separate doses of the individual mAbs (AZD8895 and then AZD1061) on Day 1.
  Interventions: Biological: AZD8895 (cell pool material); Biological: AZD1061 (cell pool material)

INTERVENTIONS:
Biological: AZD7442 — AZD7442 will be administered via IM route.
  Arms: AZD7442 (co-formulation)
Biological: AZD8895 (clonal cell line material) — AZD8895 will be administered via IM route.
  Arms: AZD8895 and AZD1061 (clonal cell line material)
Biological: AZD1061 (clonal cell line material) — AZD1061 will be administered via IM route.
  Arms: AZD8895 and AZD1061 (clonal cell line material)
Biological: AZD8895 (cell pool material) — AZD8895 will be administered via IM route.
  Arms: AZD8895 and AZD1061 (cell pool material)
Biological: AZD1061 (cell pool material) — AZD1061 will be administered via IM route.
  Arms: AZD8895 and AZD1061 (cell pool material)

SUMMARY:
The study will assess pharmacokinetic (PK) comparability between different formulations of AZD7442, which is a combination of two individual monoclonal antibodies (mAbs), AZD8895 and AZD1061.

DETAILED DESCRIPTION:
This is a randomized, open label, three-arm, single dose, parallel group, multi-center, PK comparability study.

Eligible healthy participants will be randomized in a 1:1:1 ratio between the 3 treatment groups. Each participant will receive AZD7442 as either a single intramuscular (IM) dose (co-formulation; AZD8895 + AZD1061), or as two separate IM doses of the individual mAbs (AZD8895 and then AZD1061) from either clonal cell line material or cell pool material.

Following an observation and PK and pharmacodynamic (PD) sample collection, post-dose, participants will be discharged from the Clinical Unit. During the Follow-up Period of approximately 1 year, participants will return as outpatient follow-up visits until Day 361.

The total duration of the study for a participant will be approximately 389 days comprising of a Screening Period that can last up to 28 days, Treatment Period of 1 day, and a Follow up Period of 360 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants according to medical history, physical examination, and baseline safety laboratory tests.
* Documented negative results of a Severe Acute Respiratory Syndrome Corona Virus 2 reverse transcriptase polymerase chain reaction (SARS-CoV-2 RT-PCR) test collected ≤ 3 days prior to investigational medicinal drug (IMP) dose administration (Day 1) or a negative rapid SARS-CoV-2 antigen test on Day 1 (pre-dose).
* Able to complete the Follow-up period up to Day 361 as required by the protocol.
* Body weight ≥ 50 kg to ≤ 110 kg at screening and a Body mass index ≥ 18.0 to ≤ 30 kg/m^2 at the time of the Screening Visit.

Exclusion Criteria:

* Known history of allergy or reaction to any component of AZD7442 (AZD8895 + AZD1061).
* History of infection with SARS or Middle East Respiratory Syndrome.
* Positive SARSCoV-2 result based on available data at screening or at Day 1.
* Any clinical signs and symptoms consistent with Corona virus disease 2019 (COVID-19), eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* History of clinically significant bleeding disorder.
* Active infection with hepatitis B or C or positive test for hepatitis C or for hepatitis B surface antigen at screening.
* Immunodeficiency due to illness, including HIV infection, or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone.
* Any other significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study
* Any prior receipt of another mAb indicated for the prevention or treatment of SARS CoV-2 or COVID-19.
* Receipt of a mAb within 6 months or 5 antibody half-lives.
* Receipt of a COVID-19 vaccination ≤ 14 days before IMP administration (Day 1) or plan to receive a COVID-19 vaccination ≤ 14 days after IMP dose (such participants can subsequently be included in the study once they have reached > 14 days after their last dose of vaccine).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Research Site, Anniston, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Chula Vista, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, North Hollywood, California
  - Research Site, Edgewater, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Orlando, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Berlin, New Jersey
  - Research Site, Union, South Carolina
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted_CSR_Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00009&attachmentIdentifier=fb792ba9-fb67-4ec2-948a-68d1119a8f78&fileName=D8850C00009_Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: Redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00009&attachmentIdentifier=1e4f46e2-fd37-45dc-b14d-5fa4dc023625&fileName=D8850C00009_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00009&attachmentIdentifier=8b5320ed-fd27-4bf0-aefe-ad8d9da2d0f5&fileName=D8850C00009_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 30-November-2021 (first subject first visit) to 19-July-2023 (last subject last visit).
Pre-assignment Details: A total 224 participants were randomized in this study. The screening period was up to 28 days. ICF was signed prior to screening procedures. Subjects received study drug in a randomized order. All study assessments were performed as per the schedule of assessments.
Groups:
- Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material): Participants received AZD7442 as a single intramuscular (IM) dose (co-formulation of AZD8895 + AZD1061) (clonal cell line material) on Day 1.
- Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material): Participants received AZD7442 as two separate IM doses of the individual mAbs (AZD8895 and then AZD1061) (clonal cell line material) on Day 1.
- Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material): Participants received AZD7442 as two separate IM doses of the individual mAbs (AZD8895 and then AZD1061) (cell pool material) on Day 1.
Period: Overall Study
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Started | 76 | 72 | 76
Completed | 64 | 67 | 62
Not Completed | 12 | 5 | 14
Not completed — Other | 3 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 6
Not completed — Lost to Follow-up | 4 | 1 | 7

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received any amount of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material) | Total
Number analyzed (Participants) | 76 | 72 | 76 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (14.1) | 42.4 (15.8) | 41.0 (15.2) | 42.0 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 33 | 96
  Male | 46 | 39 | 43 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 13 | 39
  Not Hispanic or Latino | 64 | 58 | 63 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 19 | 15 | 56
  White | 50 | 49 | 54 | 153
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUCinf)
Description: The pharmacokinetic (PK [AUCinf]) comparability between AZD7442 administered as a single IM dose (co-formulation) of (AZD8895 + AZD1061) versus two separate IM doses of AZD8895 followed by AZD1061: using clonal cell line material of AZD8895 and AZD1061 was evaluated. The AUCinf comparability between the clonal cell line material and the cell pool material of AZD7442 administered as two separate sequential IM doses of AZD8895 followed by AZD1061 was also evaluated.
  day*micrograms per milliliter (day*μg/mL)
Time Frame: Predose on Study Day 1 (2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose) and on Study Days 5, 8, 15, 22, 31, 61, 91, 181, 271 and 361
Population: The PK analysis set consisted of all participants in the safety analysis set who received IMP and had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure and 'number analyzed in each row' signifies the participants with available data that were analyzed for each drug for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 63 | 65 | 62
day*μg/mL
  AZD7442 | 4642 (43.12) | 4980 (38.96) | 4666 (41.06)
  AZD8895: number analyzed (Participants) | 62 | 64 | 62
  AZD8895 | 2357 (42.72) | 2634 (37.13) | 2405 (41.42)
  AZD1061 | 2326 (42.69) | 2333 (43.42) | 2255 (41.70)
Statistical Analysis 1: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUCinf of AZD7442; Test type: Other; Geometric mean ratio = 0.9380, 90% CI 2-sided [0.8458 to 1.0403]
Statistical Analysis 2: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD7442; Test type: Other; Geometric mean ratio = 0.9968, 90% CI 2-sided [0.8980 to 1.1066]
Statistical Analysis 3: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD7442; Test type: Other; Geometric mean ratio = 1.0627, 90% CI 2-sided [0.9579 to 1.1790]
Statistical Analysis 4: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUCinf of AZD8895; Test type: Other; Geometric mean ratio = 0.8992, 90% CI 2-sided [0.8107 to 0.9974]
Statistical Analysis 5: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD8895; Test type: Other; Geometric mean ratio = 0.9826, 90% CI 2-sided [0.8854 to 1.0905]
Statistical Analysis 6: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD8895; Test type: Other; Geometric mean ratio = 1.0928, 90% CI 2-sided [0.9853 to 1.2120]
Statistical Analysis 7: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUCinf of AZD1061; Test type: Other; Geometric mean ratio = 1.0039, 90% CI 2-sided [0.9029 to 1.1161]
Statistical Analysis 8: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD1061; Test type: Other; Geometric mean ratio = 1.0336, 90% CI 2-sided [0.9288 to 1.1503]
Statistical Analysis 9: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUCinf of AZD1061; Test type: Other; Geometric mean ratio = 1.0296, 90% CI 2-sided [0.9258 to 1.1451]

2. Primary Outcome: Area Under the Serum Concentration-time Curve From Day Zero to the Last Measurable Concentration (AUClast)
Description: The PK (AUClast) comparability between AZD7442 administered as a single IM dose (co-formulation) of (AZD8895 + AZD1061) versus two separate IM doses of AZD8895 followed by AZD1061: using clonal cell line material of AZD8895 and AZD1061 was evaluated. The AUClast comparability between the clonal cell line material and the cell pool material of AZD7442 administered as two separate sequential IM doses of AZD8895 followed by AZD1061 was also evaluated.
Time Frame: as for outcome 1
Population: The PK analysis set consisted of all participants in the safety analysis set who received IMP and had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 65 | 65 | 62
day*μg/mL
  AZD7442 | 4362 (43.55) | 4685 (38.60) | 4406 (40.41)
  AZD8895 | 2148 (47.37) | 2464 (36.34) | 2254 (40.54)
  AZD1061 | 2191 (43.70) | 2204 (43.62) | 2145 (41.27)
Statistical Analysis 1: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUClast of AZD7442; Test type: Other; Geometric mean ratio = 0.9418, 90% CI 2-sided [0.8512 to 1.0421]
Statistical Analysis 2: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD7442; Test type: Other; Geometric mean ratio = 0.9973, 90% CI 2-sided [0.9004 to 1.1046]
Statistical Analysis 3: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD7442; Test type: Other; Geometric mean ratio = 1.0589, 90% CI 2-sided [0.9559 to 1.1730]
Statistical Analysis 4: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUClast of AZD8895; Test type: Other; Geometric mean ratio = 0.8812, 90% CI 2-sided [0.7933 to 0.9788]
Statistical Analysis 5: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD8895; Test type: Other; Geometric mean ratio = 0.9600, 90% CI 2-sided [0.8633 to 1.0674]
Statistical Analysis 6: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD8895; Test type: Other; Geometric mean ratio = 1.0894, 90% CI 2-sided [0.9796 to 1.2116]
Statistical Analysis 7: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of AUClast of AZD1061; Test type: Other; Geometric mean ratio = 1.0065, 90% CI 2-sided [0.9061 to 1.1180]
Statistical Analysis 8: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD1061; Test type: Other; Geometric mean ratio = 1.0293, 90% CI 2-sided [0.9257 to 1.1446]
Statistical Analysis 9: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of AUClast of AZD1061; Test type: Other; Geometric mean ratio = 1.0227, 90% CI 2-sided [0.9196 to 1.1373]

3. Primary Outcome: Maximum Observed Serum (Peak) Concentration (Cmax)
Description: The PK (Cmax) comparability between AZD7442 administered as a single IM dose (co-formulation) of (AZD8895 + AZD1061) versus two separate IM doses of AZD8895 followed by AZD1061: using clonal cell line material of AZD8895 and AZD1061 was evaluated. The Cmax comparability between the clonal cell line material and the cell pool material of AZD7442 administered as two separate sequential IM doses of AZD8895 followed by AZD1061 was also evaluated.
Time Frame: as for outcome 1
Population: The PK analysis set consisted of all participants in the safety analysis set who received IMP and had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 71 | 69 | 71
Micrograms per milliliter (μg/mL)
  AZD7442 | 37.60 (40.64) | 36.48 (40.28) | 37.76 (33.64)
  AZD8895 | 18.69 (41.33) | 19.25 (37.01) | 19.37 (33.26)
  AZD1061 | 18.95 (42.15) | 17.29 (47.17) | 18.53 (36.49)
Statistical Analysis 1: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of Cmax of AZD7442; Test type: Other; Geometric mean ratio = 1.0308, 90% CI 2-sided [0.9451 to 1.1243]
Statistical Analysis 2: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD7442; Test type: Other; Geometric mean ratio = 0.9930, 90% CI 2-sided [0.9112 to 1.0822]
Statistical Analysis 3: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD7442; Test type: Other; Geometric mean ratio = 0.9634, 90% CI 2-sided [0.8833 to 1.0507]
Statistical Analysis 4: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of Cmax of AZD8895; Test type: Other; Geometric mean ratio = 0.9701, 90% CI 2-sided [0.8894 to 1.0582]
Statistical Analysis 5: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD8895; Test type: Other; Geometric mean ratio = 0.9629, 90% CI 2-sided [0.8835 to 1.0494]
Statistical Analysis 6: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD8895; Test type: Other; Geometric mean ratio = 0.9926, 90% CI 2-sided [0.9100 to 1.0826]
Statistical Analysis 7: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material); Statistical Comparison of Cmax of AZD1061; Test type: Other; Geometric mean ratio = 1.0976, 90% CI 2-sided [0.9992 to 1.2057]
Statistical Analysis 8: Comparison: Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD1061; Test type: Other; Geometric mean ratio = 1.0195, 90% CI 2-sided [0.9290 to 1.1190]
Statistical Analysis 9: Comparison: Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) vs Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material); Statistical Comparison of Cmax of AZD1061; Test type: Other; Geometric mean ratio = 0.9289, 90% CI 2-sided [0.8457 to 1.0203]

4. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax)
Description: The PK (Tmax) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Day
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 71 | 69 | 71
Day
  AZD7442 | 13.03 [2.96 to 85.01] | 14.00 [2.98 to 90.96] | 8.05 [2.97 to 61.95]
  AZD8895 | 13.02 [2.96 to 85.01] | 13.98 [2.98 to 90.96] | 8.05 [2.97 to 91.07]
  AZD1061 | 13.95 [2.96 to 55.07] | 14.00 [1.00 to 63.00] | 13.87 [2.98 to 61.95]

5. Secondary Outcome: Area Under the Serum Concentration-time Curve From Day Zero to 30 Days Post-dose (AUC0-31d)
Description: The PK (AUC0-31d) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: Study Day 1 (Predose, 2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose), and on Study Days 5, 8, 15, 22, and 31
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 70 | 67 | 68
day*μg/mL
  AZD7442 | 903.4 (44.41) | 887.9 (46.19) | 914.2 (40.53)
  AZD8895 | 447.0 (44.69) | 468.9 (42.98) | 461.7 (41.65)
  AZD1061 | 453.9 (45.65) | 415.0 (52.77) | 449.3 (42.12)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve From Day Zero to 60 Days Post-dose (AUC0-61d)
Description: The PK (AUC0-61d) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: Study Day 1 (Predose, 2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose), and on Study Days 5, 8, 15, 22, 31 and 61
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 69 | 66 | 66
day*μg/mL
  AZD7442 | 1771 (38.28) | 1752 (38.42) | 1757 (33.67)
  AZD8895 | 871.4 (39.45) | 918.9 (35.90) | 886.9 (33.87)
  AZD1061 | 894.6 (39.09) | 826.0 (43.98) | 865.8 (35.33)

7. Secondary Outcome: Area Under the Serum Concentration-time Curve From Day Zero to 90 Days Post-dose (AUC0-91d)
Description: The PK (AUC0-91d) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: Study Day 1 (Predose, 2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose), and on Study Days 5, 8, 15, 22, 31, 61 and 91
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 69 | 66 | 65
day*μg/mL
  AZD7442 | 2444 (37.20) | 2453 (36.03) | 2430 (32.95)
  AZD8895 | 1201 (38.59) | 1283 (33.67) | 1227 (32.85)
  AZD1061 | 1236 (37.94) | 1161 (41.27) | 1198 (34.51)

8. Secondary Outcome: Area Under the Serum Concentration-time Curve From Day Zero to 180 Days Post-dose (AUC0-181d)
Description: The PK (AUC0-181d) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: Study Day 1 (Predose, 2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose), and on Study Days 5, 8, 15, 22, 31, 61, 91, and 181
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 65 | 65 | 63
day*μg/mL
  AZD7442 | 3650 (39.01) | 3788 (36.10) | 3655 (36.41)
  AZD8895 | 1797 (40.54) | 1981 (33.77) | 1856 (36.27)
  AZD1061 | 1845 (39.46) | 1794 (41.11) | 1793 (37.62)

9. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast)
Description: The PK (tlast) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: Predose on Study Day 1 (2 hours, 4 hours, 8 hours post dose), Study Day 2 (24 hours post dose) and on Study Days 5, 8, 15, 22, 31, 61, 91, 181, 271 and 382
Population: as for outcome 2
Measure: Median (Full Range); unit: Day
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 65 | 65 | 62
Day
  AZD7442 | 357.98 [85.01 to 382.06] | 358.02 [60.85 to 367.97] | 357.16 [90.98 to 366.23]
  AZD8895 | 357.98 [84.99 to 382.06] | 358.02 [60.85 to 367.97] | 357.05 [90.98 to 366.23]
  AZD1061 | 357.26 [85.01 to 369.96] | 357.98 [60.85 to 367.97] | 357.16 [90.98 to 366.23]

10. Secondary Outcome: Terminal Half-life (t½λz)
Description: The PK (t½λz) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 64 | 65 | 62
Day
  AZD7442 | 75.13 (36.76) | 81.22 (29.11) | 76.52 (32.72)
  AZD8895: number analyzed (Participants) | 64 | 64 | 62
  AZD8895 | 77.77 (36.38) | 83.73 (30.12) | 79.19 (33.93)
  AZD1061 | 74.11 (34.48) | 79.19 (27.68) | 73.71 (31.06)

11. Secondary Outcome: Apparent Clearance After Extravascular Administration (CL/F)
Description: The PK (CL/F) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per day (L/day)
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 63 | 65 | 62
Liter per day (L/day)
  AZD7442 | 0.06462 (43.12) | 0.06024 (38.96) | 0.06429 (41.06)
  AZD8895: number analyzed (Participants) | 62 | 64 | 62
  AZD8895 | 0.06364 (42.72) | 0.05695 (37.13) | 0.06236 (41.42)
  AZD1061 | 0.06450 (42.69) | 0.06431 (43.42) | 0.06652 (41.70)

12. Secondary Outcome: Volume of Distribution Based on Terminal Phase After Extravascular Administration (Vz/F)
Description: The PK (Vz/F) following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs were assessed in healthy adult participants.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 63 | 65 | 62
Liter (L)
  AZD7442 | 6.960 (35.71) | 7.058 (32.17) | 7.098 (24.94)
  AZD8895: number analyzed (Participants) | 62 | 64 | 62
  AZD8895 | 7.129 (35.27) | 6.880 (30.92) | 7.125 (24.29)
  AZD1061 | 6.852 (36.99) | 7.347 (37.76) | 7.075 (26.48)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety of AZD7442 when administered as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs in healthy adult participants was assessed.
Time Frame: From Day 1 until Follow-up visit (Day 361)
Population: The safety analysis set included all participants who were randomized and received any amount of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 76 | 72 | 76
Participants
  Any AE | 21 | 21 | 26
  Any SAE | 2 | 0 | 1
  Any severe AE | 1 | 0 | 0
  Any AESI | 1 | 1 | 0
  Any SAE with outcome death | 0 | 0 | 0
  Any AE leading to study discontinuation | 0 | 0 | 0
  Any possibly related AE | 3 | 1 | 1
  Any possibly related SAE | 0 | 0 | 0
  Any possibly related severe AE | 0 | 0 | 0
  Any possibly related AESI | 1 | 1 | 0

14. Secondary Outcome: Number of Participants With Positive Anti-AZD8895 and Anti-AZD1061 Antibodies
Description: The antidrug antibody (ADA) responses to AZD7442 in serum following administration of AZD7442 as a single IM dose (co-formulation) (AZD8895 + AZD1061) and two separate IM doses (AZD8895 and then AZD1061) (clonal cell line or cell pool material) of the individual mAbs was assessed in healthy adult participants.
Time Frame: Day 1 (Pre-dose) until Follow-up visit (Day 361)
Population: The AZD8895 and AZD1061 ADA Evaluable Analysis Set included participants with at least 1 baseline and 1 post-baseline AZD8895 and AZD1061 ADA measurement. Here, 'number analyzed in each row' signifies the participants with available data that were analyzed for each drug for that outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
Number analyzed (Participants) | 73 | 70 | 71
Participants
  AZD8895: number analyzed (Participants) | 73 | 70 | 70
  AZD8895 | 6 | 2 | 2
  AZD1061 | 7 | 2 | 1

ADVERSE EVENTS:
Time Frame: From Day 1 until Follow-up visit (Day 361)
Description: The safety analysis set included all participants who were randomized and received any amount of IMP.
Arm/Group | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/72 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/76 | 0/72 | 1/76
Other Adverse Events (participants affected / at risk) | 2/76 | 8/72 | 10/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) (N=76) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) (N=72) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material) (N=76)
Major depression (Psychiatric disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: AZD8895 and AZD1061 (Coformulation, Clonal Cell Line Material) (N=76) | Treatment B: AZD8895 and AZD1061 (Separate Vials, Clonal Cell Line Material) (N=72) | Treatment C: AZD8895 and AZD1061 (Separate Vials, Cell Pool Material) (N=76)
COVID-19 (Infections and infestations) | 2 (2) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05166421/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05166421/SAP_001.pdf